CLINICAL TRIAL: NCT00531453
Title: A Phase 2, Randomized Study of VELCADE® (Bortezomib), Dexamethasone, and Thalidomide Versus VELCADE® (Bortezomib), Dexamethasone, Thalidomide, and Cyclophosphamide in Subjects With Previously Untreated Multiple Myeloma Who Are Candidates for Autologous Transplantation
Brief Title: A Study to Evaluate Two Different Regimens of VELCADE in Combination With Dexamethasone, Thalidomide and Cyclophosphamide (VDT vs VDTC) in Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-MMY-2043
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2010-06-04 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Thalidomide; Cyclophosphamide

ARMS (2):
- 1 (Experimental): bortezomib, dexamethasone, and thalidomide
  Interventions: Drug: bortezomib, dexamethasone, and thalidomide
- 2 (Experimental): bortezomib, dexamethasone, thalidomide, and cyclophosphamide
  Interventions: Drug: bortezomib, dexamethasone, thalidomide, and cyclophosphamide

INTERVENTIONS:
Drug: bortezomib, dexamethasone, and thalidomide — VELCADE (bortezomib) twice weekly for 4 cycles (4 doses per cycle), prior to high-dose chemotherapy (HDT) and stem cell transplantation(SCT). Subjects will receive VELCADE 1.3 mg/m2 as an intravenous (i.v.) bolus injection on Days 1,4,8, and 11, followed by a 10 day rest period (Days 12 to 21)
  Dexamethasone 40 mg/day will be given by mouth (p.o.) on Days 1-4 and Days 9-12 in each of 4 cycles.
  Thalidomide will be given by mouth (p.o.)every day, starting on Day 1 of Cycle 1 (e.g. the same day of the first dose of VELCADE) and continuing until Day 21 of Cycle 4 at a dose of 100 mg/day (bedtime).
  Arms: 1
Drug: bortezomib, dexamethasone, thalidomide, and cyclophosphamide — VELCADE (bortezomib) twice weekly for 4 cycles (4 doses per cycle), prior to high-dose chemotherapy(HDT)and stem cell transplantation(SCT). Subjects will receive VELCADE 1.3 mg/m2 as an intravenous (i.v.) bolus injection on Days 1,4,8, and 11, followed by a 10 day rest period (Days 12 to 21).
  Dexamethasone 40 mg/day will be given by mouth (p.o.) on Days 1-4 and Days 9-12 in each of 4 cycles.
  Thalidomide will be given by mouth (p.o.) every day, starting on Day 1 of Cycle 1 (e.g., the same day of the first dose of VELCADE) and continuing until Day 21 of Cycle 4 at a dose of 100 mg/day (bedtime).
  Cyclophosphamide will be given as an intravenous (i.v.) dose of 400 mg/m2 on Day 1 and Day 8 of each 3-week cycle, for a total of 4 cycles.
  Arms: 2

SUMMARY:
The purpose of this Phase 2 randomized study is to evaluate the efficacy and safety of treatment with a regimen of VELCADE, dexamethasone, and thalidomide (VDT) or VELCADE, dexamethasone, thalidomide, and cyclophosphamide (VDTC) in subjects with newly diagnosed symptomatic multiple myeloma who have received no prior treatment and are candidates to receive high-dose therapy and autologous bone marrow/stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between ≥18 and ≤70 years
* Patient is a candidate for HDT combined with an autologous SCT
* Karnofsky Performance Status score of ≥60%
* Multiple myeloma diagnosed according to the following standard criteria AND requiring systemic therapy:
* Presence of M-component in serum and/or urine, plus clonal plasma cells in the bone marrow and/or a documented clonal plasmacytoma
* PLUS 1 or more of the following:

  1. Calcium elevation (>11.5 mg/dL or >2.65 mmol/L)
  2. Renal insufficiency (creatinine >2 mg/dL or >177 umol/L)
  3. Anemia (hemoglobin <10 g/dL [<12.5 mmol/L] or at least 2 mg/dL [1.25 mmol/L] below normal)
  4. Bone disease (lytic lesions or osteopenia)
* AND fulfill criteria for measurable disease, as defined by at least 1 of the following 3 measurements:

  1. Serum M-protein ≥1 g/dL (≥10 g/L)
  2. Urine M-protein ≥200 mg/24 h
  3. Serum free light chain (FLC) assay: Involved FLC level ≥10 mg/dL (≥100 mg/L) provided serum FLC ratio is abnormal
* Women of childbearing potential must agree to use 2 methods of contraception.
* Males must agree to use barrier contraception.
* Subjects (or their legally acceptable representatives) must have signed an informed consent document.
* To participate in the optional pharmacogenomic component of this study, subjects (or their legally acceptable representative) must have signed the informed consent form. Refusal to consent for this component does not exclude a subject from participation in the clinical study.

Exclusion Criteria:

* Diagnosis of smoldering OR non-secretory multiple myeloma or monoclonal gammopathy of undetermined significance (MGUS).
* Diagnosis of Waldenström's disease or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
* Prior or current systemic therapy for multiple myeloma including steroids.
* Radiation therapy and/or plasmapheresis within 15 days before randomization.
* History of allergic reaction attributable to compounds being given (VELCADE, thalidomide, dexamethasone, and/or cyclophosphamide) or compounds containing boron or mannitol.
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0.
* Uncontrolled or severe cardiovascular disease
* Concurrent medical condition or disease (e.g., active systemic infection, uncontrolled diabetes) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
* Use of any investigational drugs within 30 days before randomization
* Pregnant or lactating women: A serum β-hCG pregnancy test must be performed at the Screening visit for female subjects of childbearing potential.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Wilhelminenspital-1, Vienna, Vienna, Austria

REFERENCES:
- [Result] Ludwig H; Viterbo L; Greil R; Masszi T; Spicka I; Shpilberg O; Hajek R; Dmoszynska A; Cakana A; Enny C; Feng H; van de Velde H; and Harousseau J-L. Bortezomib, Thalidomide, and Dexamethasone (VTD) Versus VTD Plus Cyclophosphamide as Induction Therapy in Previously Untreated Multiple Myeloma Patients Eligible for HDT-ASCT: A Randomized Phase 2 Trial. Blood (ASH Annual Meeting Abstracts), Nov 2009; 114: 2312.
- [Derived] Ludwig H, Greil R, Masszi T, Spicka I, Shpilberg O, Hajek R, Dmoszynska A, Paiva B, Vidriales MB, Esteves G, Stoppa AM, Robinson D Jr, Chaturvedi S, Ataman O, Enny C, Feng H, van de Velde H, Viterbo L. Bortezomib, thalidomide and dexamethasone, with or without cyclophosphamide, for patients with previously untreated multiple myeloma: 5-year follow-up. Br J Haematol. 2015 Nov;171(3):344-54. doi: 10.1111/bjh.13582. Epub 2015 Jul 7. PMID 26153365
- [Derived] Ludwig H, Viterbo L, Greil R, Masszi T, Spicka I, Shpilberg O, Hajek R, Dmoszynska A, Paiva B, Vidriales MB, Esteves G, Stoppa AM, Robinson D Jr, Ricci D, Cakana A, Enny C, Feng H, van de Velde H, Harousseau JL. Randomized phase II study of bortezomib, thalidomide, and dexamethasone with or without cyclophosphamide as induction therapy in previously untreated multiple myeloma. J Clin Oncol. 2013 Jan 10;31(2):247-55. doi: 10.1200/JCO.2011.39.5137. Epub 2012 Oct 22. PMID 23091109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 patients were enrolled between October 2007 and September 2008
Pre-assignment Details: All enrolled patients received at least one dose of study drug.
Groups:
- Three Drug Regimen (VDT): bortezomib, dexamethasone, and thalidomide
- Four Drug Regimen (VDTC): bortezomib, dexamethasone, thalidomide, and cyclophosphamide
Period: Overall Study
Arm/Group | Three Drug Regimen (VDT) | Four Drug Regimen (VDTC)
Started | 49 (02 October 2007) | 49 (02 October 2007)
Completed | 49 (10 April 2009) | 49 (10 April 2009)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Three Drug Regimen (VDT) | Four Drug Regimen (VDTC) | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 44 | 90
  >=65 years | 3 | 5 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (7.04) | 55.8 (8.27) | 55.4 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percent of Particpants Achieving Overall Combined Complete Response (CR) Following Induction
Description: Percent of Particpants Achieving Overall combined complete response (CR w/normalized serum κ:λ ratio + CR + near complete response (nCR)) following induction therapy.
  * CR criteria: negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow.
  * κ:λ ratio: normal free light chain (FLC) ratio
  * nCR criteria: positive immunofixation analysis of serum or urine as the only evidence of disease; disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow.
Time Frame: all data included in clinical database as of 10 April 2009
Population: The response-evaluable population is defined as all subjects who have measurable disease at baseline, receive at least 1 dose of any study drug and have at least 1 post-baseline response assessment. The response-evaluable population comprises 49 subjects in the VDT treatment group and 48 subjects in the VDTC group.
Measure: Number; unit: percentage of participants
Arm/Group | Three Drug Regimen (VDT) | Four Drug Regimen (VDTC)
Number analyzed (Participants) | 49 | 48
percentage of participants | 51 | 44

2. Secondary Outcome: Percent of Participants Achieving Overall Combined Complete Response (CR) Following High-dose Chemotherapy (HDT)/Stem Cell Transplantation (SCT)
Description: Percent of Participants Achieving Overall Combined Complete Response (CR) (CR w/normalized serum κ:λ ratio + CR + Near Complete Response (nCR)) following stem cell transplantation.
  * CR criteria: negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow.
  * κ:λ ratio: normal free light chain (FLC) ratio
  * nCR criteria: positive immunofixation analysis of serum or urine as the only evidence of disease; disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow.
Time Frame: all data included in clinical database as of 10 April 2009
Population: The response-evaluable population is defined as all subjects who have measurable disease at baseline, receive at least 1 dose of any study drug and have at least 1 post-transplantation response assessment. The response-evaluable population comprises 38 subjects in the VDT treatment group and 27 subjects in the VDTC group.
Measure: Number; unit: percentage of participants
Arm/Group | Three Drug Regimen (VDT) | Four Drug Regimen (VDTC)
Number analyzed (Participants) | 38 | 27
percentage of participants | 76 [NE to NE] | 78 [NE to NE]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days post last dose
Description: Treatment emergent
Arm/Group | Three Drug Regimen (VDT) | Four Drug Regimen (VDTC)
Serious Adverse Events (participants affected / at risk) | 11/49 | 20/49
Other Adverse Events (participants affected / at risk) | 48/49 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Three Drug Regimen (VDT) (N=49) | Four Drug Regimen (VDTC) (N=49)
Infections and Infestations (Infections and infestations) | 3 | 7
Gastrointestinal Disorders (Gastrointestinal disorders) | 4 | 4
General Disorders and administration site Conditions (General disorders) | 4 | 4
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 1 | 7
Respiratory, Thoracic and mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Nervous System Disorders (Nervous system disorders) | 3 | 2
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 1 | 2
Cardiac Disorders (Cardiac disorders) | 1 | 2
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 0 | 2
Metabolism and Nutritional Disorders (Metabolism and nutrition disorders) | 1 | 1
Psychiatric Disorders (Psychiatric disorders) | 0 | 1
Renal and Urinary Disorders (Renal and urinary disorders) | 1 | 0
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular Disorders (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Three Drug Regimen (VDT) (N=49) | Four Drug Regimen (VDTC) (N=49)
Gastrointestinal Disorders (Gastrointestinal disorders) | 30 | 32
General Disorders and Administration Site Conditions (General disorders) | 28 | 28
Nervous System Disorders (Nervous system disorders) | 31 | 27
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 15 | 22
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 17 | 13
Infections and Infestations (Infections and infestations) | 15 | 11
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 16 | 15
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 18 | 12
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Vascular Disorders (Vascular disorders) | 8 | 13
Psychiatric Disorders (Psychiatric disorders) | 9 | 8
Eye Disorders (Eye disorders) | 6 | 6
Hepatobiliary Disorders (Hepatobiliary disorders) | 7 | 3
Cardiac Disorders (Cardiac disorders) | 1 | 3
Investigations (Investigations) | 2 | 5
Ear and labyrinth Disorders (Ear and labyrinth disorders) | 3 | 3
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 1 | 3
Renal and Urinary Disorders (Renal and urinary disorders) | 2 | 2
Endocrine Disorders (Endocrine disorders) | 1 | 0
Immune System Disorders (Immune system disorders) | 0 | 1
Neoplasms Benign, Malignant and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Reproductive System and Brest Disorders (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No